CLINICAL TRIAL: NCT06223347
Title: A Prospective Trial Comparing Chromoendoscopy to a Digital Staining Technique and White Light in High Definition Colonoscopy in Patients With IBD Attending Scheduled Surveillance Colonoscopy
Brief Title: Improved and Simplified Staining Technique for Dysplasia Detection in Colitis
Acronym: IST-DDC
Status: Recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 281337
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Colitis; Colonic Dysplasia; Inflammatory Bowel Diseases; Colonoscopy; Surveillance
MeSH Terms: conditions — Colitis; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Chromoendoscopy — Chromoendoscopy: is a dye based staining of colonic mucosa. NBI: is an optical image enhancing technology that allows a detailed inspection of vascular and mucosal patterns, providing the ability to predict histology during real-time endoscopy.
  TXI: is a digital technique that enhance texture and color of the tissues to be more visible.
  Other Names: NBI(Narrow Band Imaging); WLI(White light); TXI( Texture and Colour Enhancement Imaging)

SUMMARY:
Comparing chromoendoscopy to a digital staining technique and White light in patients with IBD attending scheduled surveillance colonoscopy

DETAILED DESCRIPTION:
In this study we will attempt to compare dye based chromoendoscopy to WLI (white light), NBI( Narrow Band Imaging) and TXI( Texture and Colour Enhancement Imaging). High Definition Colonoscopy is used. We aim to compare all these dye/lights to each other and find the best and simplest method to help to diagnose dysplasia more efficient and easier.

ELIGIBILITY:
Inclusion Criteria:

- Person schedules to IBD- surveillance colonoscopy.

Exclusion Criteria:

* Total Colectomy.
* Not well prepared Bowel. BBPS under 2 at any segement.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Our study is directed to the IBD patients who have to undergo a surveillance colonscopy to early detection of dysplasia.
Sampling Method: Probability Sample
Enrollment: 106 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Dysplasia detection rate | 90 minutes
  Dysplasia detection rate for each staining technique

SECONDARY OUTCOMES:
Hyperplasia detection rate | 90 minutes
  Hyperplasia detection rate for each staining technique
Adenoma detection rate, ADR | 90 minutes
  Adenoma detection rate, ADR, for each staining technique
Bowel cleansing quality according to Bowel Boston Preparation Scale | 90 minutes
Serious adverse events (significant bleedings and perforations) | 90 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Molndal, Sweden

IPD SHARING:
Plan to Share IPD: No